CLINICAL TRIAL: NCT00930163
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Efficacy of Lebrikizumab (MILR1444A) in Adult Patients With Asthma Who Are Inadequately Controlled on Inhaled Corticosteroids
Brief Title: A Study of Lebrikizumab (MILR1444A) in Adult Patients With Asthma Who Are Inadequately Controlled on Inhaled Corticosteroids
Acronym: MILLY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILR4646g
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: Adult Asthma
MeSH Terms: conditions — Asthma | interventions — lebrikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: lebrikizumab (MILR1444A)
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lebrikizumab (MILR1444A) — Subcutaneous repeating dose
  Arms: 1
Drug: placebo — Subcutaneous repeating dose
  Arms: 2

SUMMARY:
This is a randomized, double-blind, placebo-controlled study to evaluate the effects of lebrikizumab in patients with asthma who remain inadequately controlled while on chronic therapy with inhaled corticosteroids (ICS).

ELIGIBILITY:
Inclusion Criteria:

* Body weight 40 kg--150 kg
* Chest radiograph with no evidence of clinically significant abnormality
* Uncontrolled asthma

Exclusion Criteria:

* Asthma exacerbation during screening
* Known malignancy
* Known immunodeficiency
* Pre-existing lung disease other than asthma
* Uncontrolled clinically significant medical disease
* Current smoker
* History of substance abuse that may impair or risk the patient's full participation in the study, in the judgment of the investigator
* Prior allergic reaction to a monoclonal antibody
* Patients (men and women) of reproductive potential who are not willing to use contraception
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change in forced expiratory volume in 1 second (FEV1) | From baseline to Week 12

SECONDARY OUTCOMES:
Change in pre-bronchodilator FEV1 | From baseline to Week 24
Change in quality of life and symptom scores | From baseline to Week 12
Change in peak flow | From baseline to Week 1
Rate of asthma exacerbations | During the 24 week treatment period
Change in rescue medication use | From baseline to Week 1
Frequency and severity of adverse events | Through study completion or early study discontinuation
Incidence of human anti-therapeutic antibodies (ATA) | At the end of the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Freemer, M.D., Study Director — Genentech, Inc.

REFERENCES:
- [Derived] Corren J, Lemanske RF, Hanania NA, Korenblat PE, Parsey MV, Arron JR, Harris JM, Scheerens H, Wu LC, Su Z, Mosesova S, Eisner MD, Bohen SP, Matthews JG. Lebrikizumab treatment in adults with asthma. N Engl J Med. 2011 Sep 22;365(12):1088-98. doi: 10.1056/NEJMoa1106469. Epub 2011 Aug 3. PMID 21812663